CLINICAL TRIAL: NCT00527605
Title: A Randomized, Double-blind, Placebo-controlled, Six-month Parallel-group Study to Assess Efficacy and Safety of Dutasteride 0.5mg Once Daily in Chinese Patients With Benign Prostatic Hyperplasia (BPH), Followed by a 12-month Open-label Treatment Phase
Brief Title: Dutasteride 0.5mg For The Treatment Of Chinese Patients With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI108898
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2011-05

CONDITIONS: Benign Prostatic Hyperplasia; Prostatic Hyperplasia
Keywords: placebo control; Chinese; Dutasteride; Randomized; Benign Prostatic Hyperplasia; Double blind
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): dutasteride 0.5mg once daily orally
  Interventions: Drug: Dutasteride 0.5mg capsule
- B (Placebo Comparator): Placebo matched once daily orally
  Interventions: Drug: Dutasteride matched placebo

INTERVENTIONS:
Drug: Dutasteride 0.5mg capsule — Dutasteride 0.5mg once daily orally
  Arms: A
Drug: Dutasteride matched placebo — Dutasteride matched placebo once daily orally
  Arms: B

SUMMARY:
This randomized, double-blind, placebo-controlled, six-month parallel-group study assess efficacy and safety of dutasteride 0.5mg once daily in Chinese patients with Benign Prostatic Hyperplasia (BPH) , followed by a 12-month open-label treatment phase

ELIGIBILITY:
Inclusion:

* Clinical diagnosis of BPH
* AUA-SI >=12 [American Urological Association Symptom Index]
* Qmax > 5ml/sec and <=15ml/sec and minimum voided volume of >=125ml
* Prostate volume >=30cm(3)

Exclusion:

* Post void residual volume >250ml
* History or evidence of prostate cancer
* Total serum PSA <1.5ng/ml or >10.0ng/ml (Prostate specific antigen)
* Previous prostatic surgery or other invasive procedures to treat BPH.
* History of AUR (Acute Urinary Retention) within 3 months
* History of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days
* Any causes other than BPH, which may in the judgement of the investigator, result in urinary symptoms or changes in flow rate
* History of hepatic impairment or abnormal liver function tests
* Use of any 5a-reductase inhibitors ,any drugs with antiandrogenic properties or other drugs noted for gynaecomastia effects, or could affect prostate volume, within past 6 months and throughout the study
* Use of alpha-receptor blockers within 2 weeks and throughout the study.
* Use of phytotherapy for BPH within 2 weeks and/or predicted to need phytotherapy during the study.
* Concurrent use of anabolic steroids
* Use of any alpha-adrenergic agonists or cholinergics within 48 hours prior to uroflowmetry assessment.
* Hypersensitivity to any 5a-reductase inhibitor or other chemically-related drugs.
* Actively trying to procreate or unwilling to wear a condom during intercourse with a woman of childbearing potential for duration of participation in this study and 16 weeks following treatment.
* History or current evidence of drug or alcohol abuse within the previous 12 months.
* History of any illness that in the opinion of the investigator might confound the results of the study or poses additional risk to the patient.
* Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, of cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of renal insufficiency, or serum creatinine >1.5xULN (Upper Limit of Normal )
* Participation in any investigational or marketed drug trial within 30 days and during the course of the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- China (7):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin

REFERENCES:
- [Background] Na Y, Ye Z, Zhang S. Efficacy and Safety of Dutasteride in Chinese Adults with Symptomatic Benign Prostatic Hyperplasia : A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study with an Open-Label Extension. Clin Drug Investig. 2012 Jan;32(1):29-39. doi: 10.2165/11593750-000000000-00000. PMID 27933597
- [Derived] Na Y, Ye Z, Zhang S; Chinese Dutasteride Phase III Trial (ARIA108898) Study Group. Efficacy and safety of dutasteride in Chinese adults with symptomatic benign prostatic hyperplasia: a randomized, double-blind, parallel-group, placebo-controlled study with an open-label extension. Clin Drug Investig. 2012 Jan 1;32(1):29-39. doi: 10.2165/11593750-000000000-00000. PMID 22017520

RESULTS

PARTICIPANT FLOW:
Groups:
- Dutasteride 0.5 mg: Oral dutasteride 0.5 milligrams (mg) once a day for 6 months
- Placebo: Matching oral placebo once a day for 6 months
Period: Overall Study
Arm/Group | Dutasteride 0.5 mg | Placebo
Started | 126 | 127
Completed | 113 | 116
Not Completed | 13 | 11
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Lost to Follow-up | 6 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride 0.5 mg | Placebo | Total
Number analyzed (Participants) | 126 | 127 | 253
Age Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.7) | 66.9 (8.2) | 66.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 126 | 127 | 253
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 126 | 127 | 253

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Prostate Volume at Month 6
Description: Percent change from baseline was calculated as the prostate volume at Month 6 minus the volume at baseline, divided by the prostate volume at baseline and multiplied by 100. Prostate volume was measured by transrectal ultrasound.
Time Frame: Baseline and Month 6
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to study treatment (after the 4-week placebo run-in) and received at least one dose of study treatment. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: percent change in volume
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 120
percent change in volume | -17.00 (21.41) | -2.77 (24.96)
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Median Difference (Final Values) = -14.23, 95% CI [-20.23 to -8.22] — Dutasteride arm minus placebo arm

2. Secondary Outcome: Percent Change From Baseline in the Prostate Volume at Month 3
Description: Percent change from baseline was calculated as the prostate volume at Month 3 minus the volume at baseline, divided by the prostate volume at baseline and multiplied by 100. Prostate volume was measured by transrectal ultrasound.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: percent change in volume
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 112 | 118
percent change in volume | -12.02 (23.22) | -1.02 (25.79)

3. Secondary Outcome: Change From Baseline in the Prostate Volume at Month 6
Description: Change from baseline was calculated as the prostate volume at Month 6 minus the volume at baseline. Prostate volume was measured by transrectal ultrasound.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 120
cubic centimeters | -9.16 (12.74) | -1.20 (12.77)

4. Secondary Outcome: Change From Baseline in the Prostate Volume at Month 3
Description: Change from baseline was calculated as the prostate volume at Month 3 minus the volume at baseline. Prostate volume is measured by transrectal ultrasound.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 112 | 118
cubic centimeters | -7.11 (13.02) | -1.06 (11.48)

5. Secondary Outcome: Percent Change From Baseline in the Serum Dihydrotestosterone (DHT) at Month 6
Description: Percent change from baseline was calculated as serum DHT at month 6 minus the value at baseline ,divided by the baseline value and multiplied by 100.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 121
percent change | -52.53 (44.42) | 26.78 (149.07)

6. Secondary Outcome: Percent Change From Baseline in the Serum DHT at Month 3
Description: Percent change from baseline was calculated as the DHT at Month 3 minus the value at baseline, divided by the baseline value and multiplied by 100.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 120
percent change | -59.15 (37.90) | 28.33 (133.71)

7. Secondary Outcome: Change From Baseline in the Serum DHT at Month 6
Description: Change from baseline was calculated as the value of DHT at Month 6 minus the baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: picograms/milliliter (pg/ml)
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 121
picograms/milliliter (pg/ml) | -289.175 (270.610) | -46.099 (399.806)

8. Secondary Outcome: Change From Baseline in the Serum DHT at Month 3
Description: Change from baseline was calculated as the value of DHT at Month 3 minus the baseline value.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 114 | 120
pg/ml | -319.605 (256.058) | -34.400 (399.633)

9. Secondary Outcome: Percent Change From Baseline in the American Urological Association Symptom Index (AUA-SI) Score at Month 6
Description: Percent change from baseline is calculated as the AUA-SI score at month 6 minus the baseline AUA-SI score, divided by the baseline score and multiplied by 100. AUA-SI is a self-administered questionnaire that assesses the severity of benign prostatic hyperplasia symptoms. Scores range from 0 to 35; mild, 0-7; moderate, 8-19; severe, 20-35.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 121
percent change | -26.48 (26.01) | -20.79 (30.18)

10. Secondary Outcome: Percent Change From Baseline in the AUA-SI Score at Month 3
Description: Percent change from baseline is calculated as the AUA-SI score at month 3 minus the baseline AUA-SI score, divided by the baseline score and multiplied by 100. AUA-SI is a self-administered questionnaire that assesses the severity of benign prostatic hyperplasia symptoms. Scores range from 0 to 35; mild, 0-7; moderate, 8-19; severe, 20-35.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 121
percent change | -15.64 (24.59) | -11.91 (21.55)

11. Secondary Outcome: Change From Baseline in the AUA-SI Score at Month 6
Description: Change from baseline was calculated as the AUS-SI score at month 6 minus the baseline score. AUA-SI is a self-administered questionnaire that assesses the severity of benign prostatic hyperplasia symptoms. Scores range from 0 to 35; mild, 0-7; moderate, 8-19; severe, 20-35.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 121
points on a scale | -4.9 (4.8) | -4.1 (5.4)

12. Secondary Outcome: Change From Baseline in the AUA-SI Score at Month 3
Description: Change from baseline was calculated as the AUA-SI score at month 3 minus the baseline score. AUA-SI is a self-administered questionnaire that assesses the severity of benign prostate hyperplasia symptoms. Scores range from 0 to 35; mild, 0-7; moderate, 8-19; severe, 20-35.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 121
points on a scale | -2.9 (3.9) | -2.4 (3.9)

13. Secondary Outcome: Percent Change From Baseline in Maximum Urinary Flow Rate (Qmax) at Month 6
Description: Percent change from baseline was calculated as Qmax at Month 6 minus Qmax at baseline, divided by baseline Qmax and multiplied by 100. Qmax is the peak urinary flow measured by a uroflow meter.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 119
percent change | 16.14 (57.43) | 6.31 (47.55)

14. Secondary Outcome: Percent Change From Baseline in Qmax at Month 3
Description: Percent change from baseline was calculated as Qmax at Month 3 minus Qmax at baseline, divided by baseline Qmax and multiplied by 100. Qmax is the peak urinary flow measured by a uroflow meter.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 111 | 117
percent change | 14.34 (42.86) | 5.85 (34.69)

15. Secondary Outcome: Change From Baseline in Qmax at Month 6
Description: Change from baseline was calculated as Qmax at Month 6 minus Qmax at baseline. Qmax is the peak urinary flow measured by a uroflow meter.
Time Frame: Baseline and Month 6
Population: ITT Population. Some participants were missing Month 6 measurements.
Measure: Mean (Standard Deviation); unit: milliliters/second (ml/s)
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 113 | 119
milliliters/second (ml/s) | 0.75 (5.61) | 0.03 (5.35)

16. Secondary Outcome: Change From Baseline in Qmax at Month 3
Description: Change from baseline was calculated as Qmax at Month 3 minus Qmax at baseline. Qmax is the peak urinary flow measured by a uroflow meter.
Time Frame: Baseline and Month 3
Population: ITT Population. Some participants were missing Month 3 measurements.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Dutasteride 0.5 mg | Placebo
Number analyzed (Participants) | 111 | 117
ml/s | 0.93 (4.74) | 0.17 (4.56)

ADVERSE EVENTS:
Time Frame: The Serious Adverse Events (SAEs) and Adverse Events (AEs) presented were collected in the 6-month Double-Blind Phase only.
Arm/Group | Dutasteride 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/126 | 1/127
Other Adverse Events (participants affected / at risk) | 27/126 | 25/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.5 mg (N=126) | Placebo (N=127)
Glaucoma (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.5 mg (N=126) | Placebo (N=127)
Palpitations (Cardiac disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 0
Pharyngitis (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 3 | 3
Throat irritation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Infections and infestations) | 0 | 1
Blood glucose increased (Infections and infestations) | 2 | 0
Prostatic specific antigen increased (Infections and infestations) | 1 | 0
White blood cell count decreased (Infections and infestations) | 1 | 0
Red blood cells urine (Infections and infestations) | 1 | 1
Transaminases increased (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Contusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Tinnitus (Nervous system disorders) | 1 | 0
Vertigo (Nervous system disorders) | 0 | 1
Poor quality sleep (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Libido decreased (Reproductive system and breast disorders) | 3 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.